CLINICAL TRIAL: NCT06833021
Title: Multicenter Retrospective Study on Hepatitis B Virus Protein X (HBx) Screening in Patients With Colitis-associated Cancer (CAC)
Brief Title: Screening for Hepatitis Virus B Protein X (HBx) in Colitis-associated Cancer (CAC)
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo (Unknown); Western University, Canada (Other)
Responsible Party: Principal Investigator, Silvio Danese, Professor, IRCCS San Raffaele
Other Study IDs: HBx-CAC
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Colitis-associated Colorectal Cancer (CAC)
Keywords: Colorectal Cancer; Hepatitis Virus B; Hepatitis Virus B Protein X; IBD; Diverticulitis; Colitis; Crohn Disease; Colitis-associated Colorectal Cancer (CAC)
MeSH Terms: conditions — Colitis-Associated Neoplasms; Colorectal Neoplasms; Diverticulitis; Colitis; Crohn Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — FFPE tissue from endoscopic biopsies or surgical resection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control Group: 33 patients used as control including patients with CRC not associated with colitis, diverticulitis, IC and CD without cancer.
  Interventions: Other: Transcriptomic Analysis
- Case Group: 33 patients diagnosed with CAC
  Interventions: Other: Transcriptomic Analysis

INTERVENTIONS:
Other: Transcriptomic Analysis — FFPE tissue blocks from patients diagnosed with CAC, including low- and high-grade dysplasia and adenocarcinoma, obtained from pathological archives will be used. RNA will be extracted and analyzed using RT-PCR to detect and quantify HBx transcripts, with Sanger sequencing employed for further validation of the results.
  Groups: Case Group
Other: Transcriptomic Analysis — RNA will be extracted and analyzed using RT-PCR to detect and quantify HBx transcripts, with Sanger sequencing employed for further validation of the results. FFPE tissue blocks from CRC, diverticulitis, IC and CD without cancer patients will be utilized as controls.
  Groups: Control Group

SUMMARY:
It was recently discovered that a protein from the Hepatitis B Virus (HBV), called HBx, is highly present in patients who were recently diagnosed with Ulcerative Colitis (UC). This was more common in UC patients than in healthy individuals or those with Crohn's Disease. About 45% of the UC patients studied had this protein, possibly due to a virus jumping from animals to humans.

In experiments with mice, it was found that HBx alone can cause colitis (inflammation of the colon) by disrupting the normal function of the gut lining. This disruption leads to inflammation and immune system problems in the colon, even without other bacteria being involved. Mice treated with HBx showed fewer immune cells, which are crucial for resolving inflammation and fighting infections. This aligns with current theories about how UC develops.

Additionally, HBx affects the genes in the gut lining, promoting cell growth and changes that could lead to cancer. In human colon tissue samples, HBx activated processes linked to the Wnt pathway, which is known to be involved in colorectal cancer. This is similar to how HBx behaves in liver cells infected with HBV, where it prevents DNA repair and leads to cancer.

Based on these findings, it is believed that HBx disrupts the balance in the gut, causing chronic inflammation that could progress to cancer. To explore this further, a study is being conducted to detect HBx in tissue samples from patients with colitis-associated cancer (CAC). Advanced techniques will be used to analyze these samples and compare them with samples from patients with other conditions like diverticulitis, indeterminate colitis, and Crohn's disease without cancer

DETAILED DESCRIPTION:
The human microbiota is a rich community of bacteria, viruses, fungi, protists, and archaea, and is an integral part of the body influencing its overall homeostasis. It colonizes all mucosal surfaces, with the gastrointestinal (GI) tract being the most densely populated. Although the most investigated gut colonizers are bacteria, emerging evidence highlights dysbiosis of the gut virome, made of both bacteriophages and eukaryotic targeting viruses, as responsible for influencing the overall intestinal microbiota composition and mucosal homeostasis by directly interacting with the other commensals, such as bacteria, or with the host, as for the eukaryotic-targeting viruses.

Eukaryotic viruses colonizing the mucosal surfaces may infect the host's cells without symptoms, and, even if asymptomatic, a virus-carrying host may hold a persistent immune response with a "continuum" of inflammatory mediators that might increase host susceptibility to disease. In parallel, eukaryotic viruses have been well-described as inducers of multiple mutational events, among which insertional mutagenesis, so viral infections are known to be responsible for about 20% of the global cancer burden. As an example, one of the most frequent infection-related cancers is hepatocarcinoma, mainly caused by the Hepatitis B virus (HBV).

Eukaryotic-targeting viruses have recently attracted considerable interest in gastrointestinal diseases such as ulcerative colitis (UC), a chronic inflammatory condition of the colonic tract, and colorectal cancer (CRC), the third most diagnosed malignancy and the fourth leading cause of cancer death in the world. UC and cancer share several factors influencing their etiogenesis, including intestinal dysbiosis. Of note, UC is a risk factor in developing colitis-associated colorectal cancer (CAC). Indeed, patients with UC have a risk of developing cancer approximately 2- to 3-fold more than the general population with poor prognosis. Dysplasia in CAC develops with different mechanisms in comparison to sporadic colorectal cancer. Patients affected by UC and CAC share a pro-inflammatory microenvironment within their mucosal tissues. Nevertheless, the mechanistic link between these two diseases is still missing.

It was recently reported that a factor derived from the Orthohepadnavirus genus, namely the Hepatitis B Virus (HBV) protein X (HBx), was the most enriched component of the virome in early-diagnosed UC patients, compared to both healthy subjects and Crohn's Disease patients. This factor was harbored by a specific cohort of UC patients (approximately 45% of the total analyzed), likely because of a zoonotic spillover event.

In vivo, HBx was shown as able to induce colitis per se independently of the other commensals, by interfering with the epithelial transcriptomic apparatus that causes the loss of appropriate barrier functions, in turn leading to the proinflammatory and immune sequelae of events within colonic mucosa, all these occurring independently of the microbiota. Indeed, HBx-treated mice displayed a reduction of neutrophils, dendritic and CD8+ T cells, indicating failure of the resolution phase (reduced neutrophils) and hampered defense against pathogens (dendritic and CD8+ T cells), all hallmarks consistent with the leading theory of UC pathogenesis. Moreover, it was shown that HBx shapes the transcriptomic state of the intestinal epithelium by binding regulatory DNA regions and activating the transcription of genes involved in the augmented epithelial cell proliferation and stemness. Notably, HBx overexpression in human colonic mucosa biopsies induced activation of biological processes related to the Wnt pathway, which is involved in colorectal carcinogenesis. This result is consistent with the HBx description in the context of HBV infection. Indeed, this viral protein is known to prevent the HBV-infected hepatocytes from efficiently repairing damaged DNA, thus leading to an accumulation of DNA mutations and, eventually, hepatocarcinogenesis.

Based on this evidence and preliminary results, it is believed that HBx-mediated epithelial alterations affect mucosal homeostasis, disrupting and driving intestinal chronic inflammation, which may progress to dysplastic lesions or adenocarcinoma.

For this reason, a multicenter retrospective study is being conducted to investigate the presence of HBx in patient-derived samples from individuals diagnosed with CAC. In detail, the study will employ reverse transcription polymerase chain reaction (RT-PCR) and Sanger sequencing techniques to analyze Formalin-Fixed Paraffin-Embedded (FFPE) tissue samples to detect HBx. A control group will be included, comprising CRC samples from patients without colitis and samples from patients with diverticulitis, indeterminate colitis (IC), and Crohn's disease (CD) without cancer.

The assessment of HBx in CAC samples could revolutionize clinical approaches by enabling earlier diagnosis and refining risk assessment for patients with UC. This finding may also lead to the development of personalized treatment strategies that specifically target HBx-related pathways, thereby advancing the understanding of the underlying disease mechanisms

ELIGIBILITY:
Inclusion Criteria:

* adult patients (age ≥18 years), both male and female, diagnosed with CAC, CRC, diverticulitis, IC or CD who had previously undergone endoscopic biopsy or surgical resection, according to standard clinical practice (from 2021 to 2024);
* patients with no documented history of HBV infection;
* patients who had already signed the informed consent authorizing the use of their clinical data for future scientific research.

Exclusion Criteria:

* patients under 18 years of age;
* adult patients (age ≥18 years), both male and female diagnosed with CAC, CRC, diverticulitis, IC or CD with a documented history of HBV infection;
* patients who have not signed the informed consent authorizing the use of their clinical data for future scientific research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 66 total patients, of which 33 diagnosed with CAC and 33 representing the control group composed of CRC without colitis, diverticulitis, and CD without cancer. 20 patients will be enrolled at our center, and the remaining 40 will be equally distributed among the participating units: IRCCS Casa Sollievo della Sofferenza Hospital (San Giovanni Rotondo (FG), Italy) and Western University (London, Ontario, Canada).
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
To define HBx as a predictive biomarker of CAC in UC patients | Being a retrospective study, we plan to collect FFPE stored from October 2021 to December 2024. Duration of total study period: 12 months.
  FFPE tissue blocks from patients diagnosed with CAC, including low- and high-grade dysplasia and adenocarcinoma, obtained from pathological archives will be used. RNA will be extracted and analyzed using RT-PCR to detect and quantify HBx transcripts, with Sanger sequencing employed for further validation of the results. Additionally, FFPE tissue blocks from CRC, diverticulitis, IC and CD without cancer patients will be utilized as controls. FFPE tissue blocks already present in the Pathology Unit will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Silvio Danese, PhD-MD, Study Director — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided